CLINICAL TRIAL: NCT06836986
Title: COMPARISON BETWEEN EFFICACY OF NOREPINEPHRINE AND PHENYLEPHRINE BOLUSES FOR PREVENTION OF SPINAL ANAESTHESIA INDUCED HYPOTENSION IN OBSTETRICAL PATIENTS UNDERGOING EMERGENCY CESAREAN SECTION- A Double Blind Randomized Controlled Trial
Brief Title: COMPARISON BETWEEN EFFICACY OF NOREPINEPHRINE AND PHENYLEPHRINE BOLUSES for PREVENTION OF SPINAL ANAESTHESIA INDUCED HYPOTENSION IN OBSTETRICAL PATIENTS UNDERGOING EMERGENCY CESAREAN SECTION-A Double Blind Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Rabia Kamal, FCPS Anesthesiology resident, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: spinal induced hypotension
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Spinal Anesthesia Induced Hypotension
Keywords: Spinal anesthesia induced hypotension; Emergency lower segment cesarean section; Norepinephrine bolus; Prophylactic; Phenylephrine

STUDY DESIGN:
Intervention Model Description: This study has two groups of participants. Group N and group P. Allocation of participants in each group is being done by basic randomization.
Who Masked: Participant, Investigator
Masking Description: both participants and investigator is unaware about the drug given. Data is being collected by the anesthesiologist who is not involved in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group P (Active Comparator): Prophylactic bolus of phenylephrine will be administered right after spinal anesthesia induction
  Interventions: Drug: Phenylephrine bolus
- Group N (Experimental): Prophylactic bolus of norepinephrine will be administered right after spinal anesthesia.
  Interventions: Drug: Norepinephrine Bolus

INTERVENTIONS:
Drug: Norepinephrine Bolus — Prophylactic norepinephrine bolus of 8 micrograms will be administered right after spinal anesthesia induction.
  Rescue bolus of norepinephrine 4 micrograms will be administered in case of hypotension.
  Arms: Group N
Drug: Phenylephrine bolus — Prophylactic phenylephrine bolus of 100 micrograms will be administered right after spinal anesthesia induction.
  Rescue bolus of phenylephrine 50 micrograms will be administered in case of hypotension.
  Arms: Group P

SUMMARY:
The goal of this clinical trial is to learn if norepinephrine is more effective than phenylephrine for prevention of spinal anesthesia induced hypotension. The main questions it aims to answer are:

Does norepinephrine lower the incidence of spinal anesthesia induced hypotension in emergency obstetrical patients? We will compare effectiveness of norepinephrine and phenylephrine for the prevention of spinal anesthesia induced hypotension.

Participants will:

Be administered prophylactic boluses of both drugs right after spinal anesthesia induction and maternal hemodynamic parameters and neonatal APGAR scores will be recorded

DETAILED DESCRIPTION:
Spinal anesthesia is a common mode of anesthesia in cesarean delivery. Spinal anesthesia induced hypotension is one of the most common complication that can affect both mother and fetus. For the management of spinal anesthesia induced hypotension, preloading with crystalloids and colloids, use on ionotropic agents and vasopressors have already been in practice.

Objective of this study is to compare efficacy of prophylactic use of norepinephrine and phenylephrine bolus dosage for spinal anesthesia induced hypotension.

This study is being conducted at the department of anesthesiology ,K.M Pfau civil hospital, Dow university of health sciences, Karachi , Pakistan. Data is being collected after taking approval from Institutional review board and written informed consent from the participants.

Participants are being enrolled by primary investigator. All participants are undergoing simple randomization by lottery method.

After enrollment of participants, demographic data, hemodynamic parameters and other relevant details are being recorded till delivery of the neonate.

Hemodynamic parameters that are heart rate, systolic and diastolic blood pressure, mean arterial blood pressure is being recorded every 3mins. APGAR scoring of neonate is also being recorded.

After completion of data collection, data will be done using Statistical package for social sciences 26.

ELIGIBILITY:
Inclusion Criteria:

1. American society of anesthesiologists II and III patients
2. Age 18-40years
3. Gestational age 32 weeks and above

Exclusion Criteria:

1. Patients with hypertensive disorders of pregnancy having baseline systolic blood pressure greater than 160 mmHg and diastolic blood pressure greater than 99 mmHg.
2. Baseline mean arterial pressure less than 70 mmHg.
3. Antepartum hemorrhage/intraoperative blood loss greater than 1000ml
4. history indicative of cardiovascular or neurological disease.
5. known fetal abnormality.
6. Patients taking serotonin reuptake inhibitor, Tricyclic antidepressants,monoamine oxidase inhibitors.
7. Maternal situations requiring immediate administration of general anesthesia

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 124 (Estimated)
Dates: Start 2024-12-31 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of spinal anesthesia induced Hypotension | From induction of spinal anesthesia till delivery of neonate
  Prophylactic norepinephrine and phenylephrine boluses will be administered to both groups right after spinal anesthesia induction.greater than 80% drop of the Systolic blood pressure will be defined as hypotension.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Ruth km pfau civil hospital karachi Dow University of health sciences, department of anesthesiology, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
participants confidentiality

REFERENCES:
- [Background] Nadella H, Islam A, Ina EA, Levin D, Bacoat-Jones T. The Management of Spinal and Epidural Anesthesia-Related Hypotension in the United States During Cesarean Childbirth. Cureus. 2024 Mar 17;16(3):e56340. doi: 10.7759/cureus.56340. eCollection 2024 Mar. PMID 38633922
- [Background] Ng K, Parsons J, Cyna AM, Middleton P. Spinal versus epidural anaesthesia for caesarean section. Cochrane Database Syst Rev. 2004;2004(2):CD003765. doi: 10.1002/14651858.CD003765.pub2. PMID 15106218